CLINICAL TRIAL: NCT00249002
Title: A Pilot Phase II Trial Of ABI-007 (A Cremophor El-Free, Protein Stabilized, Nanoparticle Paclitaxel) For The Prevention Of Vascular Access Graft Failure In Patients Undergoing Hemodialysis
Brief Title: Use of ABI-007 for the Prevention of Vascular Access Graft Failure in Patients Undergoing Hemodialysis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to pipeline prioritization
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HD001
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Hemodialysis Graft Dysfunction
Keywords: Vascular Access Graft Failure; Venous Neointimal Hyperplasia(VNH); Hemodialysis
MeSH Terms: interventions — Albumin-Bound Paclitaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABI-007 (Experimental): ABI-007 35 mg/m^2 given intravenously (IV) into the arteriovenous (AV) graft within 96 hours after angioplasty, followed by repeat treatment during weeks 5, 13 and 21
  Interventions: Drug: ABI-007

INTERVENTIONS:
Drug: ABI-007
  Other Names: Abraxane®; paclitaxel

SUMMARY:
This study is designed to confirm the safety of the proposed dose and schedule of ABI-007 for hemodialysis patients with vascular access device failure, and to obtain preliminary data on the effectiveness of such treatment.

DETAILED DESCRIPTION:
This is an open-label, pilot, phase II study to assess the feasibility of administering ABI-007 intravenously [IV] over 3-5 minutes to patients with hemodialysis graft dysfunction (i.e., either a thrombosed polytetrafluoroethylene (PTFE) graft, or a patent but dysfunctional PTFE graft). Patients with graft dysfunction who are successfully treated with angioplasty will start treatment after angioplasty or during their first dialysis through the graft following intervention, and will receive 3 subsequent treatments of ABI-007 at 35 mg/m^2 on weeks 5, 13 and 21.

ELIGIBILITY:
Inclusion Criteria:

* Thrombosed graft within the past 7 days or a patent but dysfunctional polytetrafluoroethylene (PTFE) graft (identified by any means) with a stenosis of greater than 50% at the graft-vein anastomosis or within 8 centimeters of the graft-vein anastomosis which will be referred to as the index lesion. Following angioplasty patients must have residual stenosis of less than 20% post angioplasty for the index lesion and for all other stenoses; also index lesion must be located in the arm. PTFE graft requiring angioplasty must be at least 30 days old.
* Male or non-pregnant and non-lactating female, and ≥ 18 years of age.
* Patient or guardian has provided a signed written informed consent for the administration of ABI-007 (post-angioplasty or at the time of first dialysis through the new graft) using a form that is approved by the local IRB/ethics committee of the investigative site.
* Patient or his/her legally authorized representative or guardian has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent form prior to participation in any study-related activities.

Exclusion Criteria:

* Use of a stent at the time of current angioplasty or at any previous time in the index lesion.
* No perforation at the time of current angioplasty.
* Thrombosed graft for more than 7 days.
* Patient has the following blood counts at baseline:
* Absolute neutrophil count (ANC) < 2.0*10^9/L;
* platelets < 100*10^9/L;
* Hemoglobin (Hgb) < 9 g/dL.
* Patient has the following blood chemistry levels at baseline:
* Aspartate transaminase (AST or SGOT), alanine transaminase (ALT or SGPT) > 2.5x upper limit of normal range (ULN);
* total bilirubin ≥ upper limit of normal (ULN);
* Unable to give informed consent, or for whom informed consent cannot be obtained from a legal guardian.
* Women who are pregnant and women of child bearing potential who do not use adequate contraception.
* 2 procedures of percutaneous or surgical intervention on the PTFE graft within the previous 90 days.
* Previous participation in another study with any investigational drug or device within the past 30 days or current enrollment in any other clinical protocol or investigational trial.
* Patient has a life expectancy of less than 6 months.
* Intended kidney transplant within 6 months of enrollment in the study
* Any significant medical condition which in the investigators opinion may interfere with the patients optimal participation in the study.
* Patient is, in the investigator's opinion, unlikely to be able to complete the study through the End of Study (EOS) visit.
* Patient has a history of allergy or hypersensitivity to the study drug.
* Documented hypercoagulable state requiring anti-coagulation (protein S, protein C, antiphospholipid; anticoagulation on an empiric basis for graft thromboses in not a contradiction).
* Patient is human immunodeficiency virus (HIV) positive.
* Patient is currently receiving other chemotherapy drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-11-01 (Actual); Primary Completion 2007-11-01 (Actual); Study Completion 2007-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Iglesias, MD, Study Director — Celgene Corporation
Locations (4):
- United States (4):
  - Peoria, Illinois
  - Shreveport, Louisiana
  - Rochester, New York
  - Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABI-007
Started | 9
Completed | 2
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Study cancellation | 3
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | ABI-007
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (8.16)
Age, Customized [Number; unit: participants]
  <65 years | 4
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black of African heritage | 7
  White, Non-Hispanic and Non-Latino | 2
  White, Hispanic or Latino | 0
  Other | 0
Weight [Mean (Standard Deviation); unit: kg] | 71.78 (13.271)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Discontinued, Delayed or Interrupted Therapy
Description: Percentage of participants who had discontinued therapy or had a delayed dose or an interrupted (omitted) dose due to toxicities/adverse events.
Time Frame: up to week 21
Population: Treated population
Measure: Number; unit: percentage of participants
Arm/Group | ABI-007
Number analyzed (Participants) | 9
percentage of participants
  Delayed dose | 44
  Interrupted | 0
  Discontinued therapy | 33

2. Primary Outcome: Percentage of Participants Without Graft Failure or Need for Intervention
Description: Graft failure is defined as graft thrombosis, loss of vascular access function, or >50% stenosis of the index lesion at the time of a regularly scheduled angiographic assessment.
Time Frame: 24 weeks
Population: Evaluable participants who were treated
Measure: Number; unit: percentage of participants
Arm/Group | ABI-007
Number analyzed (Participants) | 7
percentage of participants | 0

3. Primary Outcome: Stenosis (%) of the Index Lesion at Venous Anastomosis Using Angiography at Week 12
Description: Indexed lesion must be located in the arm and is a polytetrafluoroethylene (PTFE) thrombosed graft or a patent but dysfunctional PTFE graft with a residual stenosis of less than 30% after the pre-dose angioplasty. The percent of stenosis (narrowing) of the index lesion is measured by angiography.
Time Frame: 12 weeks
Population: Treated population of participants with an index lesion at this site.
Measure: Mean (Standard Deviation); unit: percentage of stenosis
Arm/Group | ABI-007
Number analyzed (Participants) | 6
percentage of stenosis | 61.7 (32.51)

4. Primary Outcome: Stenosis (%) of the Index Lesion at Venous Anastomosis Using Angiography at Week 24
Description: as for outcome 3
Time Frame: 24 weeks
Population: Treated population of participants with an index lesion at this site.
Measure: Mean (Standard Deviation); unit: percentage of stenosis
Arm/Group | ABI-007
Number analyzed (Participants) | 5
percentage of stenosis | 79.0 (11.40)

5. Secondary Outcome: Participants With Arthrosclerotic Cardiovascular Complications
Description: Counts of participants who had treatment-emergent arthrosclerotic cardiovascular complications, specifically myocardial infarction, arterial thromboses, or cerebrovascular events.
Time Frame: up to week 25
Population: Treated population
Measure: Number; unit: participants
Arm/Group | ABI-007
Number analyzed (Participants) | 9
participants
  >=1 arthrosclerotic cardiovascular complication | 4
  Bradycardia | 1
  Hypotension | 1
  Hypertrophic obstructive cardiomyopathy | 1
  Carotid artery stenosis | 1
  Cerebrovascular accident | 1
  Cardiovascular disorder | 1

6. Secondary Outcome: Kaplan Meier Estimates for Time to Graft Failure or Intervention
Description: The time to graft failure or intervention was defined as the time from first dose of study drug to the first time graft failure or intervention. Participants who did not have graft failure or intervention at the end of the study were censored at the last known time that the participant had angiography.
Time Frame: up to 12 months
Population: Treated population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | ABI-007
Number analyzed (Participants) | 8
weeks | 11.4 [11.0 to 12.0]

7. Secondary Outcome: Percentage of Participants With Patency of Index and Non-Index Lesions at 24 Weeks
Description: The patency (unblocking) for index lesions is defined as <50% of stenosis and no PFTE graft thrombosis at 24 weeks. The patency for non-index lesions is defined as <50% of stenosis and no new non-index lesions at 24 weeks.
Time Frame: 24 weeks
Population: Treated Population of evaluable participants
Measure: Number; unit: percentage of participants
Arm/Group | ABI-007
Number analyzed (Participants) | 7
percentage of participants
  Index lesion | 14
  Non-Index lesions | 57

8. Primary Outcome: Stenosis (%) of the Index Lesion at Venous Anastomosis Using Angiography at Month 9
Description: as for outcome 3
Time Frame: 9 months
Population: Treated population of participants with an index lesion at this site.
Measure: Mean (Standard Deviation); unit: percentage of stenosis
Arm/Group | ABI-007
Number analyzed (Participants) | 3
percentage of stenosis | 69.3 (4.04)

9. Primary Outcome: Stenosis (%) of the Index Lesion at Venous Anastomosis Using Angiography at Month 12
Description: as for outcome 3
Time Frame: 12 months
Population: Treated population of participants with an index lesion at this site.
Measure: Number; unit: percentage of stenosis
Arm/Group | ABI-007
Number analyzed (Participants) | 1
percentage of stenosis | 95.0

10. Primary Outcome: Stenosis (%) of a Non-index Lesion Using Angiography at Week 12
Description: Non-indexed lesion with a residual stenosis of less than 30% after the pre-dose angioplasty. The percent of stenosis (narrowing) of the non-index lesion is measured by angiography. Three non-index lesions are reported: central vein, intragraft and arterial anastomosis.
Time Frame: 12 weeks
Population: Treated population of participants with a non-index lesion.
Measure: Mean (Standard Deviation); unit: percentage of stenosis
Arm/Group | ABI-007
Number analyzed (Participants) | 2
percentage of stenosis
  Central vein | 50.0 (NA) — only one participant
  Intragraft | 35.0 (35.36)
  Arterial anastomosis | 25.0 (NA) — only one participant

11. Primary Outcome: Stenosis (%) of a Non-index Lesion Using Angiography at Week 24
Description: as for outcome 10
Time Frame: 24 weeks
Population: Treated population of participants with a non-index lesion.
Measure: Mean (Standard Deviation); unit: percentage of stenosis
Arm/Group | ABI-007
Number analyzed (Participants) | 2
percentage of stenosis
  Central vein | 40.0 (NA) — only one participant
  Intragraft | 45.0 (21.21)
  Arterial anastomosis | 27.5 (NA) — only one participant

12. Primary Outcome: Stenosis (%) of a Non-index Lesion Using Angiography at Month 9
Description: as for outcome 10
Time Frame: 9 months
Population: Treated population of participants with a non-index lesion.
Measure: Mean (Standard Deviation); unit: percentage of stenosis
Arm/Group | ABI-007
Number analyzed (Participants) | 2
percentage of stenosis
  Central vein | 65.0 (NA) — only one participant
  Intragraft | 57.5 (10.61)
  Arterial anastomosis | 25.0 (NA) — only one participant

13. Primary Outcome: Stenosis (%) of a Non-index Lesion Using Angiography at Month 12
Description: as for outcome 10
Time Frame: 12 months
Population: Treated population of participants with a non-index lesion.
Measure: Number; unit: percentage of stenosis
Arm/Group | ABI-007
Number analyzed (Participants) | 1
percentage of stenosis
  Central vein | NA (NA) — no participants at this timepoint
  Intragraft | 50.0
  Arterial anastomosis | 25.0

ADVERSE EVENTS:
Time Frame: AEs collected up to 30 days after the last ABI-007 dose administration (Week 21), except for cardiovascular side effects or other events at the investigator's discretion, which would be reported whenever they occur.
Arm/Group | ABI-007
Serious Adverse Events (participants affected / at risk) | 6/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-007 (N=9)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 2 (2)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-007 (N=9)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 3 (4)
Vascular graft complication (Injury, poisoning and procedural complications) | 2 (4)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (2)
Hypertrophic obstructive cardiomyopathy (Cardiac disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Facial palsy (Nervous system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Study data will not be published in part before the complete multicenter data has been reported in full, unless more than 1 year has elapsed since completion of the Study.
* Investigator/institution must supply copy of presentation or publication to Celgene within 30 days of submission for publication. Celgene may request in writing within that 30 days that Celgene Confidential Information be deleted or be granted a 60 day delay prior to publication to permit intellectual property filings.